CLINICAL TRIAL: NCT06912230
Title: Appetite and Energy Intake in Young Female Adults During and After Simulated High-Altitude
Brief Title: Hypoxia, Appetite, and Energy Intake in Young Female Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); Hopital Montfort (Other); Institut du Savoir Montfort (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H-06-18-837
Record Dates: First submitted 2025-03-17; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-10

CONDITIONS: Hypoxia; Altitude; Appetite; Energy Intake
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normoxia (Experimental)
  Interventions: Other: Normoxia
- Hypoxia (simulated altitude of 5000 meters above sea-level) (Experimental)
  Interventions: Other: Hypoxia (simulated altitude of 5000 meters above sea-level)

INTERVENTIONS:
Other: Normoxia — Participants will undergo a 6-hour passive exposure to normoxia in a climate-controlled environmental chamber maintained at 22°C with 30% relative humidity. They will remain in a fasted state throughout the exposure period.
  Arms: Normoxia
Other: Hypoxia (simulated altitude of 5000 meters above sea-level) — Participants will undergo a 6-hour passive exposure to a simulated altitude of 5000 meters above sea-level in a climate-controlled environmental chamber maintained at 22°C with 30% relative humidity. They will remain in a fasted state throughout the exposure period.
  Arms: Hypoxia (simulated altitude of 5000 meters above sea-level)

SUMMARY:
The goal of this clinical trial is to investigate the effects of acute passive continuous hypoxemia (simulated high-altitude at rest) on appetite and energy intake in healthy young female adults. The main questions it aims to answer are:

* Does six hours of simulated high-altitude (5000 meters) reduce scores of subjective appetite and energy intake?
* Do changes in appetite and energy intake persist in the hours following the end of hypoxic exposure? Researchers will compare the effects of simulated high-altitude to a control normoxia (sea-level) condition to see if exposure to low oxygen levels independently affect appetite and energy intake.

Participants will:

* Visit the laboratory for a preliminary screening session to assess eligibility.
* Undergo two randomized, single-blind, experimental sessions consisting of six hours of passive exposure to normoxia or hypoxia in a climate-controlled chamber.
* Consume foods provided from a curated list, served in ad libitum quantities, after leaving the laboratory to assess post-exposure energy intake.

ELIGIBILITY:
Inclusion Criteria:

* English or French speaking
* Ability to provide informed consent

Exclusion Criteria:

* History or evidence of chronic disease
* Current use of hypolipemic medication
* Current use of hormonal contraceptives
* Current use of antidepressants
* Current use of anticoagulants
* Ongoing smoking status
* Experiencing pregnancy, puerperium, or irregular menstrual cycles

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in desire to eat | Baseline and 6 hours; Baseline and 24 hours
  Scores of subjective desire to eat, measured using visual analog scales. Measurements are performed upon arrival at the laboratory (baseline), hourly during the exposure, immediately after a 30-minute ad libitum buffet, immediately before bedtime, and 24 hours after the baseline measurement.
Change from baseline in hunger | Baseline and 6 hours; Baseline and 24 hours
  Scores of subjective hunger, measured using visual analog scales. Measurements are performed upon arrival at the laboratory (baseline), hourly during the exposure, immediately after a 30-minute ad libitum buffet, immediately before bedtime, and 24 hours after the baseline measurement.
Change from baseline in fullness | Baseline and 6 hours; Baseline and 24 hours
  Scores of subjective fullness, measured using visual analog scales. Measurements are performed upon arrival at the laboratory (baseline), hourly during the exposure, immediately after a 30-minute ad libitum buffet, immediately before bedtime, and 24 hours after the baseline measurement.
Change from baseline in prospective food consumption | Baseline and 6 hours; Baseline and 24 hours
  Scores of subjective prospective food consumption, measured using visual analog scales. Measurements are performed upon arrival at the laboratory (baseline), hourly during the exposure, immediately after a 30-minute ad libitum buffet, immediately before bedtime, and 24 hours after the baseline measurement.
Energy intake immediately after 6 hours of exposure (buffet) | Hour 6 of exposure
  Energy intake in the laboratory during a 30-minute ad libitum buffet immediately after 6 hours of exposure, administered using a validated food menu (McNeil, 2012) and analyzed using the Food Processor SQL from ESHA Research, Inc.
Energy intake post-buffet | 6.5 hours of exposure and 24 hours
  Energy intake outside the laboratory between end-buffet and bedtime, administered using a validated food menu (McNeil, 2012) and analyzed using the Food Processor SQL from ESHA Research, Inc.

SECONDARY OUTCOMES:
Heart rate | 6 hours
  Measured continuously throughout the exposure.
Oxyhemoglobin saturation | 6 hours
  Measured continuously throughout the exposure.
Systolic blood pressure | 6 hours
  Measured upon arrival at the laboratory (baseline), hourly during the exposure, and immediately after eating.
Diastolic blood pressure | 6 hours
  Measured upon arrival at the laboratory (baseline), hourly during the exposure, and immediately after eating.
Lake Louise Acute Mountain Sickness Score | 6 hours
  Peak score on the Lake Louise Acute Mountain Sickness questionnaire, measured upon arrival at the laboratory (baseline), hourly during the exposure, and immediately after eating.
Fluid consumption during exposure | 6 hours
  Average hourly fluid consumption calculated by weighing participant water intake at the start and end of each hour of exposure (normalized to the exposure duration).
Fluid loss during exposure | 6 hours
  Fluid loss calculated as the change in body mass during each exposure presented as a percentage of baseline body mass (corrected for fluid consumption)
Change from baseline in explicit liking using the LFPQ | Baseline and 6.5 hours of exposure
  Explicit liking will be measured using the Leeds Food Preference Questionnaire. Measurements will be taken upon arrival at the laboratory (baseline), following 5 hours of exposure, and after a 30-min ad libitum buffet.
Change from baseline in explicit wanting using the LFPQ | Baseline and 6.5 hours of exposure
  Explicit wanting will be measured using the Leeds Food Preference Questionnaire. Measurements will be taken upon arrival at the laboratory (baseline), following 5 hours of exposure, and after a 30-min ad libitum buffet.
Change from baseline in implicit wanting using the LFPQ | Baseline and 6.5 hours of exposure
  Implicit wanting will be measured using the Leeds Food Preference Questionnaire. Measurements will be taken upon arrival at the laboratory (baseline), following 5 hours of exposure, and after a 30-min ad libitum buffet.
Change from baseline in olfaction | Baseline and Hour 4 of exposure
  Olfaction will be measured using the Sniffin' Sticks (Burghart Instruments, Wedel, Germany), a 3-test battery of odorized markers that measure odor detection threshold, odor discrimination, and odor identification. Measurements will be performed upon arrival at the laboratory (baseline) and following 4 hours of exposure.
Change from baseline in gustation | Baseline and Hour 4 of exposure
  Olfaction will be measured using Taste Strips (Burghart Instruments, Wedel, Germany). Measurements will be performed upon arrival at the laboratory (baseline) and following 4 hours of exposure.
Change from baseline in resting energy expenditure | Baseline and Hour 5 of exposure
  Resting energy expenditure will be measured via indirect calorimetry upon arrival at the laboratory (baseline) and following 5 hours of exposure.
Change from baseline in respiratory exchange ratio | Baseline and Hour 5 of exposure
  Respiratory exchange ratio will be measured via indirect calorimetry upon arrival at the laboratory (baseline) and following 5 hours of exposure.
Change from baseline in plasma glucose concentrations | 6 hours
  Plasma glucose concentrations will be measured via colorimetric assays from venous blood samples collected upon arrival at the laboratory (baseline) and hourly during the exposure (i.e., 0 or baseline, 60, 120, 180, 240, 300, and 360 minutes).
Change from baseline in plasma insulin concentrations | 6 hours
  Plasma insulin concentrations will be measured via colorimetric assays from venous blood samples collected upon arrival at the laboratory (baseline) and hourly during the exposure (i.e., 0 or baseline, 60, 120, 180, 240, 300, and 360 minutes).
Change from baseline in plasma non-esterified fatty acid concentrations | 6 hours
  Plasma non-esterified fatty acid concentrations will be measured via colorimetric assays from venous blood samples collected upon arrival at the laboratory (baseline) and hourly during the exposure (i.e., 0 or baseline, 60, 120, 180, 240, 300, and 360 minutes).
Change from baseline in plasma triglyceride concentrations | 6 hours
  Plasma triglyceride concentrations will be measured via colorimetric assays from venous blood samples collected upon arrival at the laboratory (baseline) and hourly during the exposure (i.e., 0 or baseline, 60, 120, 180, 240, 300, and 360 minutes).
Change from baseline in plasma beta-hydroxybutyrate concentrations | 6 hours
  Plasma beta-hydroxybutyrate concentrations will be measured via colorimetric assays from venous blood samples collected upon arrival at the laboratory (baseline) and hourly during the exposure (i.e., 0 or baseline, 60, 120, 180, 240, 300, and 360 minutes).

CONTACTS AND LOCATIONS:
Locations (1):
- Behavioural and Metabolic Research Unit, School of Human Kinetics, Faculty of Health Sciences, University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No